CLINICAL TRIAL: NCT00076544
Title: An Open-Label, Long-Term, Multi-Center, Intrathecal Ziconotide (PRIALT) Effectiveness and Safety Trial (ZEST) in Patients With Chronic Severe Pain
Brief Title: Ziconotide Effectiveness and Safety Trial in Patients With Chronic Severe Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Elan Pharmaceuticals (Industry)
Allocation: Non-Randomized | Masking: None | Purpose: Treatment
Other Study IDs: ELN92045-501
Record Dates: First submitted 2004-01-26; First posted 2004-02-04 (Estimated); Last update posted 2015-12-14 (Estimated); Status verified 2015-12

CONDITIONS: Pain
Keywords: Intrathecal
MeSH Terms: conditions — Pain | interventions — ziconotide

INTERVENTIONS:
Drug: Ziconotide

SUMMARY:
The purpose of this open-label study is to give chronic severe pain patients with existing intrathecal pump systems access to ziconotide.

ELIGIBILITY:
Inclusion Criteria:

* Each patient must have chronic severe pain of malignant or nonmalignant etiology with inadequate pain relief from or intolerance to conventional therapy.
* Each patient must have a predicted life expectancy of greater than or equal to 6 weeks relative to baseline.
* Each patient must be able to respond to the Visual Analog Scale of Pain Intensity (VASPI).
* Each patient must have an implanted programmable SynchroMed infusion device or a CADD-Micro external programmable infusion device and spinal catheter (hereafter "IT pump and spinal catheter") prior to enrollment into this trial. (If a patient has an external pump, the Investigator must ensure that the patient is at a low risk for infection and that the patient is capable of maintaining good personal hygiene. The Investigator must have demonstrated the ability to successfully manage patients with external pumps prior to enrolling a patient in this trial.)
* Each patient must be at least 18 years of age.
* Each patient must be competent to give written informed consent and has given written informed consent prior to performance of any study-related procedures. Reasonable accommodation of visually impaired patients will be allowed.
* Each patient is willing and able to comply with the protocol requirements.
* Each female patient of childbearing potential must agree to use adequate contraceptive methods while on PRIALT as determined by the Investigator.

Exclusion Criteria:

* Presence of pregnancy or lactation.
* Participation in another investigational drug or device trial within the preceding 30 days.
* Presence of known hypersensitivity to PRIALT or any of its components.
* Presence of any contraindication to continued IT therapy (for example, infection at the pump or catheter externalization site, uncontrolled bleeding diathesis, spinal canal obstruction that impairs cerebrospinal fluid [CSF] circulation, or patient and caregiver inability to manage and protect the IT pump and spinal catheter system and return for clinic follow up visits).
* Presence of any condition (for example, psychosis, severe depression or suicidal ideation, homicidality, somatization disorder, active substance abuse, cognitive deficits, dementia or other serious medical or psychiatric condition) that in the Investigator's opinion precludes the patient's ability to participate in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300
Dates: Start 2004-02; Primary Completion 2005-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (65):
- United States (65):
  - Alabama Pain Center, Huntsville, Alabama
  - Center for Pain Management, Huntsville, Alabama
  - Otto Uhrik, MD, Sun City West, Arizona
  - Outcomes Research International, Tucson, Arizona
  - The RC Goodman Pain Institute, Fort Smith, Arkansas
  - Innovative Spine Care, Little Rock, Arkansas
  - Shreenath Clinical Services, Beverly Hills, California
  - Advanced Pain Institute, Duarte, California
  - Shreenath Clinical Services, Lake Forest, California
  - Shreenath Clinical Services, Long Beach, California
  - Bay Area Pain Center, Los Gatos, California
  - Northridge Surgery & Pain Management Center, Northridge, California
  - Pacific Pain Medicine Consultants, Oceanside, California
  - Pacific Pain Treatment Centers, San Francisco, California
  - Galileo Surgery Center, San Luis Obispo, California
  - Pain Relief Center of Colorado, Arvada, Colorado
  - Pain Care Specialists, Colorado Springs, Colorado
  - Rocky Mountain Clinical Research, Golden, Colorado
  - Comprehensive Pain and Headache Treatment Centers, LLC, Derby, Connecticut
  - Florida Institute of Medical Research, Jacksonville, Florida
  - Space Coast Pain Institute, Merritt Island, Florida
  - West Gables Rehabilitation Hospital, Miami, Florida
  - Sarasota Pain Associates, Sarasota, Florida
  - Clinical Pharmacology Services, Tampa, Florida
  - Shepherd Center, Inc., Atlanta, Georgia
  - Comprehensive Pain Care, PC, Marietta, Georgia
  - The University of Chicago, Dept. of Surgery, Section of Neurosurgery, Chicago, Illinois
  - Indianapolis Neurosurgical Group, Indianapolis, Indiana
  - University of Iowa Health Care, Iowa City, Iowa
  - Des Moines Orthopedic Surgeons, West Des Moines, Iowa
  - University of Kentucky, Lexington, Kentucky
  - Pain Control Network, PSC/PCN Surgical Suites, LLC, Louisville, Kentucky
  - Wayne State University - School of Medicine, Detroit, Michigan
  - Medical Advanced Pain Specialists (MAPS), Minneapolis, Minnesota
  - The Center for Pain Medicine, Hattiesburg, Mississippi
  - Pain Management Associates, Clinical Research, Independence, Missouri
  - St. John's Regional Healthcare, Springfield, Missouri
  - Pain Management - Anesthesiology, Las Vegas, Nevada
  - Dr. O'Connell's Pain Care Centers, Inc., Somersworth, New Hampshire
  - All Island Pain Consultants, Bay Shore, New York
  - Cohn Pain Management Center, Bethpage, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - NYU Pain Management Center, New York, New York
  - New York Presbyterian Hospital/Cornell Medical Center, New York, New York
  - Medical Pain Management of Central New York, Syracuse, New York
  - Duke Medical Center Pain Clinic, Durham, North Carolina
  - The Center for Clinical Research, Winston-Salem, North Carolina
  - Cincinnati Centers for Pain Relief, Inc., Hamilton, Ohio
  - PETC Research Group, Inc., Tulsa, Oklahoma
  - Pain Consultants of Oregon, Eugene, Oregon
  - Pain Management Consultants, PC, Portland, Oregon
  - Lehigh Valley Hospital, Allentown, Pennsylvania
  - Magee Rehabilitation, Philadelphia, Pennsylvania
  - Carolinas Center for Advanced Management of Pain, Spartanburg, South Carolina
  - Avera St. Luke's Hospital, Aberdeen, South Dakota
  - Dallas Spine Care P.A., Dallas, Texas
  - Advanced Pain Medicine, Dallas, Texas
  - The University of Texas Medical Branch, Galveston, Texas
  - International Pain Institute, Lubbock, Texas
  - American Pain & Wellness, PA, Plano, Texas
  - Consultants in Pain Research, PA, San Antonio, Texas
  - Lifetree Clinical Research, Salt Lake City, Utah
  - University of Utah Pain Management Center, Salt Lake City, Utah
  - Pain Management Center, University of Virginia, Charlottesville, Virginia
  - The Center for Pain Relief, Charleston, West Virginia